CLINICAL TRIAL: NCT02695927
Title: Rehabilitation Glasses for the Treatment of Hemispatial Neglect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chun Lim (Other)
Responsible Party: Sponsor-Investigator, Chun Lim, Physician, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009P000297
Record Dates: First submitted 2015-09-07; First posted 2016-03-01 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: 1/2 patients receive visual stimulation with rehabilitation glasses. 1/2 patients receive control stimulation with rehabilitation glasses.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chronic (Experimental): Crossover study on the benefits of computer rehabilitation glasses on chronic sufferers of hemispatial neglect
  Interventions: Device: Computer rehabilitation glasses
- Acute (Experimental): Randomized, controlled study on the benefits of computer rehabilitation glasses on acute sufferers of hemispatial neglect
  Interventions: Device: Computer rehabilitation glasses
- Optimization (Experimental): Study to identify optimal operating parameters of computer rehabilitation glasses
  Interventions: Device: Computer rehabilitation glasses
- Duration (Active Comparator): Study to determine duration of effect of computer rehabilitation glasses
  Interventions: Device: Computer rehabilitation glasses

INTERVENTIONS:
Device: Computer rehabilitation glasses

SUMMARY:
This project is designed to test a lightweight, portable, computerized pair of glasses that will help reduce some of the cognitive deficits seen in patients who have suffered damage to their right cerebral hemisphere.

DETAILED DESCRIPTION:
Hemispatial neglect is the inability or failure to attend and respond to the left side of space. Patients suffering right cerebral hemispheric damage from stroke or traumatic brain injury frequently suffer neglect and will ignore all information located in the left side of space. Currently there is no effective rehabilitation technique to treat neglect and many of these patients have severe long-term disability. The goal of this project is to determine whether a prototypical pair of rehabilitation glasses can reduce the symptoms of hemispatial neglect.

ELIGIBILITY:
Inclusion Criteria:

* Presence of hemispatial neglect as defined by Behavioral Inattention Test score of 129 or worse (maximum score 146).

Exclusion Criteria:

* Presence of aphasia at time of testing,
* Recent seizures
* Major psychiatric illness
* Prior unrelated neurological disease

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-03; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Improvement of patient's hemispatial neglect scores | 60 days
  Behavioral Inattention Test

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon publication of the data. Other researchers can contact PI to request this data.

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963